CLINICAL TRIAL: NCT05999266
Title: The Effect of Ultrasonographic Cartilage Thickness and Quadriceps/Hamstring Muscle Thickness on Knee Pain in Patients With Rheumatoid Arthritis
Brief Title: The Cartilage and Muscle Thickness on Knee Pain in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 15082023
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis; Knee Pain Chronic; Muscle Loss; Cartilage Degeneration
MeSH Terms: conditions — Arthritis, Rheumatoid; Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis Patients with Knee Pain: In patients with knee pain, the cartilage thickness measurement of the knee joint will be measured from 3 points by ultrasound. At the same time, Quadriceps and Hamstring muscle thickness measurements of the patients will be made from the midpoints where the muscle thickness is the highest.
  Interventions: Diagnostic Test: Ultrasonographic Measurements
- Rheumatoid Arthritis Patients without Knee Pain: In patients without knee pain, the cartilage thickness measurement of the knee joint will be measured from 3 points by ultrasound. At the same time, Quadriceps and Hamstring muscle thickness measurements of the patients will be made from the midpoints where the muscle thickness is the highest.
  Interventions: Diagnostic Test: Ultrasonographic Measurements

INTERVENTIONS:
Diagnostic Test: Ultrasonographic Measurements — In patients with or without knee pain, the cartilage thickness measurement of the knee joint will be measured from 3 points by ultrasound. At the same time, Quadriceps and Hamstring muscle thickness measurements of the patients will be made from the midpoints where the muscle thickness is the highest.

SUMMARY:
The knee pain status of the patients who are followed in the rheumatology special branch of the Physical Medicine and Rehabilitation Outpatient Clinic and who meet the inclusion criteria will be questioned. In patients with or without knee pain, the cartilage thickness measurement of the knee joint will be measured from 3 points by ultrasound. At the same time, Quadriceps and Hamstring muscle thickness measurements of the patients will be made from the midpoints where the muscle thickness is the highest. The physician who performed the ultrasonographic measurements of the knee pain status of the patients does not know.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis > Diagnosed for 1 year
* -Female gender
* -The patient has been in remission or low disease activity for at least 3 months
* -Be able to ambulatory
* -No significant deformity in the lower extremity joints

Exclusion Criteria:

* Patient with active arthritis or high disease activity

  * - Significant deformity of the lower extremity joints and inability to ambulate
  * -Pregnant patient
  * - Presence of malignancy
  * - Patient with a severe psychiatric disorder and difficulty in cooperation
  * - Presence of cardiovascular and pulmonary comorbidities that will prevent exercise
  * -Male gender

Ages: 30 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with Rheumatoid Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Cartilage Thickness Measurement | through study completion, an average of 1 month
  Tibial cartilage thickness will be visualized by ultrasound with the knee held in 30 degrees of flexion, and 3 measurements will be taken from the medial, lateral and midline.
Ultrasonographic Muscle Measurement Thickness Measurement | through study completion, an average of 1 month
  The quadriceps muscle thickness will be measured by determining the midpoint between the SIAS and the patella while the patient is lying in the supine position. Hamstring muscle thickness will be measured at the intersection of a line drawn at 60% distal between the greater trochanter and the outer femoral condyle, and at the midline of the popliteal fossa, with the patient lying on the prone. These 2 measurements will be proportional to each other.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)